CLINICAL TRIAL: NCT05929144
Title: Optimization of MRI Sequences Used in the Study of Neurodegenerative Diseases at Inserm U1237 NeuroPresage Team, Cyceron Center in Caen
Brief Title: Optimization of MRI Sequences Used in the Study of Neurodegenerative Diseases
Acronym: IRMtests
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0030; 2023-A00398-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2023-05-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other)
  Interventions: Other: MRI sequences testing

INTERVENTIONS:
Other: MRI sequences testing — Testing different MRI sequences in order to optimize them

SUMMARY:
The Inserm NeuroPresage team has been using MRI for more than 20 years in the study of normal ageing and memory pathologies to further the understanding and the characterization of early diagnosis and the cerebral substrates of cognitive deficits in patients, particularly in the context of neurodegenerative diseases.

Two years ago, a new 3T MRI camera was installed at the Cyceron centre. It is more efficient and should make it possible to obtain better quality images and/or to reduce the time required to acquire these images.

In this context, it seems important to test the different sequences that we classically use in our studies, or that we plan to implement in our next studies (learning and text retrieval fMRI task), in order to optimize them, with a view to integrating them in our future studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of legal age
* Affiliation with a social security scheme or beneficiary of such a scheme
* Signing of the protocol informed consent
* For women of childbearing age or capacity, a urine pregnancy test before inclusion

Exclusion Criteria:

* Protected persons in accordance with articles L. 1121-5 to L.1121-8 of the Public Health Code: protected adults, pregnant and nursing women
* Presence of contraindications to MRI examination without contrast agents injection
* Presence of a chronic neurological or psychiatric condition (including substance use disorder)
* History of brain disease (vascular, degenerative, malformative, tumour, or head trauma with loss of consciousness for more than one hour)
* Current or recent use of medications that may interfere with imaging (psychotropic drugs, antihistamines with anticholinergic action, antiparkinsonian drugs, benzodiazepines including muscle relaxants, long-term steroidal anti-inflammatory drugs, antiepileptic drugs, central painkillers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Optimization of MRI sequences | During MRI sessions
  TR, TE, Flip Angle, asset phase, asset slice parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gaël Chételat, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Nicolas Cabé, MD, PhD, Principal Investigator — CHU Caen Normandie
Locations (1):
- GIP Cyceron, Caen, France

IPD SHARING:
Plan to Share IPD: No